CLINICAL TRIAL: NCT04769193
Title: A Clinical Trial Evaluating the Efficacy of a Skin Cream Targeting Dermal Fat in Improving the Skin Elasticity of Healthy Volunteers
Brief Title: A Clinical Trial Evaluating the Efficacy of a Skin Cream in Improving Facial Appearance and Skin Elasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adipeau Inc. (Industry)
Collaborators: Romo Plastic Surgery (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adipeau-001
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Atrophy, Hemifacial; Elastosis; Photoaging
Keywords: Sagging; Depletion; Atrophy; Photoaging
MeSH Terms: conditions — Facial Hemiatrophy; Atrophy

STUDY DESIGN:
Masking Description: The evaluation of skin volume will be masked as the assessors will not known which scans are from what time period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adipeau face cream (Experimental): Cosmetic cream
  Interventions: Other: Adipeau face cream

INTERVENTIONS:
Other: Adipeau face cream — Adipeau face cream contains the natural actives Carthamus Tinctorius (Safflower) Seed Oil and Kaempferia Parviflora Rhizome Extract (Black Ginger).

SUMMARY:
A Clinical Trial Evaluating Efficacy of a Skin Cream Targeting Dermal Fat in Improving the Skin Elasticity of Healthy Volunteers.

DETAILED DESCRIPTION:
This is a single-arm study with subjects serving as their own controls. The study evaluates a face cream comprised of natural agents with adipogenic and lipolytic activities. The combination of adipogenic and lipolytic impulses is theorized to be more effective in promoting regeneration and healthy cell size in the dermal white adipose tissue than other approaches (e.g., adipogenic + lipogenic or anti-adipogenic + lipolytic). The health of the dermal white adipose tissue is reflected by the strength and elasticity of the skin and the distribution of volume in the face.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Plans to undergo facial skin resurfacing (e.g. laser, chemical peel, microneedling) during the study period
* Plans to undergo injectable filler treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-03-27 (Estimated); Study Completion 2022-06-27 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Elasticity | Six months and 12 months..
  Elasticity measured by DermaLab Skin Elasticity Meter.
Change in Skin Volume | Six months and 12 Months.
  Increases and decreases measured by Cherry Imaging 3D Scanning System.

SECONDARY OUTCOMES:
FaceQ skin satisfaction surveys | Two, Six and 12 Months.
  Satisfaction With Skin, Appraisal of Lower Eyelids, Satisfaction with Cheeks, Adverse Effects

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Tower, MD, Principal Investigator — Romo Plastic Surgery
Locations (1):
- Thomas Romo Plastic Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galanin I, Nicu C, Tower JI. Facial Fat Fitness: A New Paradigm to Understand Facial Aging and Aesthetics. Aesthetic Plast Surg. 2021 Feb;45(1):151-163. doi: 10.1007/s00266-020-01933-6. Epub 2020 Sep 10. PMID 32914326